CLINICAL TRIAL: NCT03272243
Title: Short Segment Posterior Fixation With Index Level Screws Versus Long Segment Posterior Fixation for Thoracolumbar Spine Fracture: Angle of Correction and Pain
Brief Title: Short Segment vs Long Segment Fixation in Traumatic Dorsolumbar Spine Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Nada, Fellow of functional neurosurgery division, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G10800
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: SPINAL Fracture
Keywords: thoracolumbar fracture; short segment fixation; long segment fixation; index level
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Segment posterior spine fixation (Active Comparator): Short segment transpedicular screw fixation with inclusion of the index level
  Interventions: Procedure: short segment posterior spine fixation
- Long Segment posterior spine fixation (Active Comparator): Long segment transpedicular screw fixation with escape of the index level
  Interventions: Procedure: long segment posterior spine fixation

INTERVENTIONS:
Procedure: short segment posterior spine fixation
  Arms: Short Segment posterior spine fixation
Procedure: long segment posterior spine fixation
  Arms: Long Segment posterior spine fixation

SUMMARY:
A prospective study included 91 patients, who had single level thoracolumbar fracture with Cobb's angle ≤ 25⁰, underwent posterior fixation. Forty four patients underwent short segment fixation with screws into the index level, and 47 patients underwent long segment fixation with skipped index level. The angle of correction, pain, and neurological state were regularly assessed

ELIGIBILITY:
Inclusion Criteria:

* wedge fracture or burst fracture with Thoraco-Lumbar Injury Classification and Severity (TLICS) score ≥ 4
* Single level fracture
* Less than 50% of spinal canal compromised
* Mild kyphosis or scoliosis
* Cobb's angle ≤ 25˚
* with or without neurological deficit

Exclusion Criteria:

* patients with multiple level fractures
* patients with more than 50% spinal canal compromise
* patients who needed anterior approach to decompress the canal
* patients who have fracture dislocation and / or marked kyphosis and scoliosis with Cobb's angle >25⁰
* patients who needed 360⁰ fixation with long segment fixation to maintain the angle of correction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change in pain | 3rd, 6th, 9th, 12th months
  Visual analogue scale assessment
Change in disability | 3rd, 6th, 9th, 12th months
  assessment of Oswestry Disability Scale
Change in angle of correction | 3rd, 6th, 9th, 12th months
  Measurement of Cobb's angle

CONTACTS AND LOCATIONS:
Overall Officials: Walid A Abdel Ghany, M.D., Ph.D, Study Director — Associate Professor of Neurosurgery

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR